CLINICAL TRIAL: NCT06457646
Title: mRNA Expression and Genetic Polymorphisms Affecting DRD3 (rs6280) and HTR2A (rs6313) in Bruxism
Status: Not yet recruiting | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Yosra Gassara, Principal Investigator, University of Monastir
Other Study IDs: 011/2021; 0000-0002-5945-7764 (Other: 0000-0002-5945-7764)
Record Dates: First submitted 2024-06-01; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Bruxism
Keywords: Gene Expression; Bruxism; Sleep bruxism; Polymorphism; Genetic
MeSH Terms: conditions — Bruxism; Sleep Bruxism | interventions — Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Genetic: Genetic polymorphism — The biological significance of HTR2A and DRD3 in bruxism remains unclear as molecular analyses, including genetic association studies, have not explored the mRNA expression of genes implicated in bruxism. This study aims to evaluate the influence of genetic polymorphisms affecting DRD3 (rs6280) and HTR2A (rs6313) on bruxism to identify potentially associated genotypes. Additionally, it aims to investigate the expression of HTR2A and DRD3 to elucidate their biological significance in bruxism.

SUMMARY:
The goal of this observational study is to learn about the genetic factors influencing bruxism, a condition characterized by teeth grinding, in a group of participants. The main questions it aims to answer are:

* Is there a significant association between the rs6313 polymorphism of the HTR2A gene and bruxism?
* Is there a significant association between the rs6280 polymorphism of the DRD3 gene and bruxism?

Participants will:

Provide DNA samples for genotyping of the DRD3 (rs6280) and HTR2A (rs6313) polymorphisms.

Provide RNA samples to assess changes in the expression of HTR2A and DRD3. Researchers will compare the genetic data and RNA expression levels between individuals with bruxism and those without (controls) to see if there are significant genetic differences and expression changes associated with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* be above 18 years of age and have a confirmed diagnosis of bruxism

Exclusion Criteria:

* Systemic diseases,
* orofacial dysfunction,
* acute symptoms such as neurodegenerative diseases (specifically Parkinsons disease),
* Taking medication such as anxiolytics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 170 participants will be included in this study.
Sampling Method: Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2024-06-02 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
PCR-RFLP Analysis | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wieckiewicz M, Bogunia-Kubik K, Mazur G, Danel D, Smardz J, Wojakowska A, Poreba R, Dratwa M, Chaszczewska-Markowska M, Winocur E, Emodi-Perlman A, Martynowicz H. Genetic basis of sleep bruxism and sleep apnea-response to a medical puzzle. Sci Rep. 2020 May 4;10(1):7497. doi: 10.1038/s41598-020-64615-y. PMID 32367059
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32367059/